CLINICAL TRIAL: NCT06581315
Title: Efficacy and Safety of Donafenib as Adjuvant Therapy for Postoperative Patients With High-Risk Recurrent Hepatocellular Carcinoma: A Multicenter, Randomized Controlled Study
Brief Title: Postoperative Adjuvant Therapy of Donafenib for Hepatocellular Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYXKY-2024-666-02
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Hepatocellular Carcinoma; Adjuvant Therapy
Keywords: Hepatocellular Carcinoma; Adjuvant Therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — donafenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Donafenib) (Experimental): Participants will receive Donafenib treatment until disease recurrence or unacceptable toxicity or up to 1 years.
  Interventions: Drug: Donafenib
- Arm B (active surveillance) (No Intervention): Active surveillance of participants.

INTERVENTIONS:
Drug: Donafenib — Donafenib 100 mg twice daily (BID)
  Other Names: Zepsun
  Arms: Arm A (Donafenib)

SUMMARY:
This study aims to evaluate the efficacy and safety of donafenib as adjuvant therapy for postoperative patients with high-risk recurrent Hepatocellular Carcinoma. This is a multicenter, randomized controlled study.

ELIGIBILITY:
Inclusion Criteria:

* Participants underwent radical resection of hepatocellular carcinoma 4 weeks before randomization
* High Risk of recurrence as assessed by tumor characteristics
* Without any anti-tumor therapy before surgery, except preoperative TACE therapy, traditional Chinese medicine therapy and interferon therapy
* Child-Pugh Class A statu
* ECOG Performance Status of 0 or 1
* CT/MR confirmed no recurrence or metastasis at ≥4 weeks after surgery
* Expected survival time of no less than 3 months

Exclusion Criteria:

* Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC
* Evidence of residual or a history of spontaneous tumor rupture
* Recurrent HCC
* Prior received Liver transplantation
* Prior anti tumor therapy for treatment of HCC (including sorafenib or any other molecular therapy, anti-PD-1 antibody and other immunotherapies, FOLFOX systemic chemotherapy) is excluded
* AFP does not return to normal 4 weeks after operation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2024-08-28 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2032-08-30 (Estimated)

PRIMARY OUTCOMES:
One year recurrence-free survival (RFS) rate | 1 year
  The proportion from randomization to 1 year without recurrence.

SECONDARY OUTCOMES:
Recurrence-Free Survival (RFS ) | 6 years
  The time from randomization to disease recurrence, or death from any cause (whichever occurs first).
Recurrence-Free Survival rate (RFS rate) | 5 years
  The proportion from randomization to 2 years, 3 years or 5 years without recurrence.
Overall Survival (OS) | 6 years
  The time from randomization to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Changzhen Shang, MD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No